CLINICAL TRIAL: NCT03438617
Title: Peer Support To Enhance The Shanghai Integration Model Of Diabetes Care: Extension & Dissemination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai 6th People's Hospital (Other)
Collaborators: University of North Carolina, Chapel Hill (Other); Asian Center for Health Education (Other); Shanghai Municipal Commission of Health and Family Planning (Other)
Responsible Party: Principal Investigator, Weiping Jia, Professor, Director of Shanghai Institute of Diabetes, Shanghai Sixth People's Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai 6th People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-197
Record Dates: First submitted 2018-01-24; First posted 2018-02-20 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes; Self-Management; Primary Care; Community Health Center; Peer Support; Group Support; Integrated Care; China; Urban
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Original Design: This study uses a stepped wedge design in three successive cohorts. Ten community health centers (CHC) will be randomized to one of three cohorts, 3 CHCs in the first cohort vs. 3 CHCs in the second cohort vs. 4 CHCs in the third cohort.
  Actual Implementation: The Peer Leader program was designed as an implementation study to assess the feasibility, effectiveness and sustainability of integrating peer support with routine care in CHCs. 10 CHCs were selected in this community-based prospective cohort study according to their having in place the key organizational resources and willingness to collaborate. However, one CHC withdrew due to its administrator's judgement of insufficient staff resources for implementation, resulting in 9 CHCs. A planned, stepped wedge design to stagger introduction of the program over subsets of CHCs proved impractical within the realities of those sites. Finally, 9 CHCs participated in this study as one single interventional group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Peer Support Intervention (Experimental): 9 CHCs will receive the peer support intervention for the full duration of the study period (12 months). Baseline assessment, 12-month and 18-month evaluation to assess the effectiveness and sustainability of the intervention.
  Interventions: Behavioral: Peer Support

INTERVENTIONS:
Behavioral: Peer Support — The intervention involves monthly education/support groups co-led by a CHC doctor / nurse and peer leaders. These meetings will begin with a general discussion about participants' previous month, what they had been doing, any special events etc. Meetings will devote time to identifying goals and specific plans for reaching them, rehearsal and/or discussion of specific behaviors to execute plans and ways in which the group members can be helpful to each other. This will be organized around a Diabetes Action Plan. Peer leaders will also organize activities to promote healthy lifestyles, such as walking groups, to promote informal contacts among peer leaders and participants.

SUMMARY:
This project developed a combined model of the Shanghai Integration Model and peer support for diabetes self-management education and support. The program was implemented and evaluated in nine Community Health Centers in Shanghai, China.

Note: This registration reflects modifications to a study that was registered in 2018.

DETAILED DESCRIPTION:
The development of contemporary diabetes care offers new hope for long and satisfying lives of those with the disease, but also provides increased challenges for integration across the many dimensions of care (varied medications in addition to insulin, specialty services, diet, physical activity, stress management, etc.) and across the many who contribute to care (specialists, primary care providers, nurses, dietitians and patient educators, family members, friends, worksites). The Shanghai Integration Model (SIM) has made great strides to integrating specialty/hospital care with primary/community care. The addition of peer support can enhance patient engagement within that integrated care. Peer support can also integrate care with the daily behaviors and patterns that optimal diabetes management requires and with the family members and others in individuals' daily lives who can support diabetes management.

This project developed a combined model of the Shanghai Integration Model and peer support for diabetes self-management education and support. The program was implemented and evaluated in nine Community Health Centers (CHCs) in Shanghai, China. The program is a collaboration among the Shanghai Sixth People's Hospital, Shanghai Jiao Tong University, the Shanghai Diabetes Institute, the Shanghai Health Bureau, the Shanghai Centers for Disease Control, and, at the University of North Carolina-Chapel Hill, Peers for Progress, widely recognized for its leadership in promoting peer support in health care and prevention.

A planned, stepped wedge design to stagger introduction of the program over subsets of CHCs proved impractical within the realities of those sites. Therefore, the original study protocol was modified in the following ways:

* Instead of staggering program implementation among 3 cohorts of CHCs, all participating CHCs implemented the program concurrently in a single-arm design.
* A greater number of participants were enrolled than anticipated.
* To reduce risk of Type 1 error, the number of secondary endpoints was reduced to those central to diabetes management - glycemia, blood pressure, and lipids, and, in the area of psychosocial factors, depression, diabetes distress, and general quality of life.
* The original plan called for outcome measures to be collected at baseline, 3 months, 6 months, and 12 months according to the stepped wedge study design. Since the CHCs implemented the program in one cohort, the outcome measures were collected at baseline, 12 months, and 18 months in order to assess the long term benefits given the chronic, progressive nature of diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Chinese
* Has type 2 diabetes
* Receiving treatment at participating community health center

Exclusion Criteria:

* Severe mental illness (severe depression, schizophrenia, bipolar disorder, obsessive compulsive disorder, panic disorder, PTSD, borderline personality disorder, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1284 (Actual)
Dates: Start 2017-03-08 (Actual); Primary Completion 2019-02-11 (Actual); Study Completion 2019-02-11 (Actual)

PRIMARY OUTCOMES:
Change from Baseline HbA1c at 12 and 18 months | Baseline, 12 months, 18 months
  HbA1c (%)

SECONDARY OUTCOMES:
Change from Baseline Blood Pressure at 12 and 18 months | Baseline, 12 months, 18 months
  SBP and DBP (mmHg)
Change from Baseline Blood Lipids at 12 and 18 months | Baseline, 12 months, 18 months
  LDL (mmol/L)
Change from Baseline General Quality of Life at 12 and 18 months | Baseline, 12 months, 18 months
  5-item measure of quality of life adapted from the EQ-5D, a standardized instrument for measuring generic health status. The respondents are asked to choose one of the statements which best describes their health status on the surveyed day. Rated level can be coded as a number 1, 2, or 3, which indicates having no problems for 1, having some problems for 2, and having extreme problems for 3. As a result, a person's health status can be defined by a 5-digit number, ranging from 11111 (having no problems in all dimensions) to 33333 (having extreme problems in all dimensions). A sixth item, the visual analogue scale, was not included.
Change from Baseline Diabetes Distress at 12 and 18 months | Baseline, 12 months, 18 months
  4-item measure of diabetes distress adapted from the 17-item Diabetes Distress Scale. The respondents are asked to respond to which degree each of the items has bothered them in the past month on a 6-point scale (1-6), where 1 is not a brother and 6 is very bothersome. Scores are summed and divided by 4 to calculate the mean.
Change from Baseline Depression at 12 and 18 months | Baseline, 12 months, 18 months
  8-item Patient Health Questionnaire (PHQ), the PHQ-9 minus the last question on suicidal thoughts. The PHQ is a standard instrument used in primary care settings to screen for the presence and severity of depression. The respondents are asked how often they have been bothered by each of the 8 items in the past 2 weeks on a 4 point scale (0-3), where 0 is "not all" and 3 is "nearly every day". The scores for each item are summed to produce a total score between 0 and 24 points. A total score of 0 to 4 represents no significant depressive symptoms. A total score of 5 to 9 represents mild depressive symptoms; 10 to 14, moderate; 15 to 19, moderately severe; and 20 to 24, severe.

CONTACTS AND LOCATIONS:
Overall Officials: Weiping Jia, MD, PhD, Principal Investigator — Shanghai 6th People's Hospital; Edwin B Fisher, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (10):
- China (10):
  - Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality
  - An Ting Community Health Center, Shanghai, Shanghai Municipality
  - Cao Yang Community Health Center, Shanghai, Shanghai Municipality
  - Hong Mei Community Health Center, Shanghai, Shanghai Municipality
  - Kang Jian Community Health Center, Shanghai, Shanghai Municipality
  - Long Hua Community Health Center, Shanghai, Shanghai Municipality
  - Nan Jing Xi Road Community Health Center, Shanghai, Shanghai Municipality
  - Tao Pu Community Health Center, Shanghai, Shanghai Municipality
  - Tian Lin Community Health Center, Shanghai, Shanghai Municipality
  - Zhen Ru Community Health Center, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fisher EB, Boothroyd RI, Coufal MM, Baumann LC, Mbanya JC, Rotheram-Borus MJ, Sanguanprasit B, Tanasugarn C. Peer support for self-management of diabetes improved outcomes in international settings. Health Aff (Millwood). 2012 Jan;31(1):130-9. doi: 10.1377/hlthaff.2011.0914. PMID 22232103
- [Background] Zhong X, Wang Z, Fisher EB, Tanasugarn C. Peer Support for Diabetes Management in Primary Care and Community Settings in Anhui Province, China. Ann Fam Med. 2015 Aug;13 Suppl 1(Suppl 1):S50-8. doi: 10.1370/afm.1799. PMID 26304972
- [Background] Chan JC, Sui Y, Oldenburg B, Zhang Y, Chung HH, Goggins W, Au S, Brown N, Ozaki R, Wong RY, Ko GT, Fisher E; JADE and PEARL Project Team. Effects of telephone-based peer support in patients with type 2 diabetes mellitus receiving integrated care: a randomized clinical trial. JAMA Intern Med. 2014 Jun;174(6):972-81. doi: 10.1001/jamainternmed.2014.655. PMID 24781960